CLINICAL TRIAL: NCT02204124
Title: Thunderbeat™ Integrated Bipolar and Ultrasonic Forceps in the Whipple Procedure: A Prospective Registry Trial
Brief Title: Whipple Procedure: Standard of Care vs. Thunderbeat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator and Study Sponsor decided to terminate the study early
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201311146
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Neoplasms; Bile Duct Carcinoma
Keywords: Whipple procedure
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Ligation; Surgical Instruments; Sutures

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be blinded to the assigned operating technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Active Comparator): In the control group, scissors, ligatures, clips and sutures will be used for dissection and hemostasis as necessary.
  Interventions: Device: Standard of care scissors, ligatures, clips, and sutures
- Thunderbeat™ (Experimental): -In the Thunderbeat™ group, dissection and hemostasis of vessels will be performed using the Thunderbeat™ device (Olympus, Japan).
  Interventions: Device: Thunderbeat

INTERVENTIONS:
Device: Thunderbeat — Thunderbeat uses ultrasonic and high frequency bipolar energy simultaneously to seal and cut tissue compared to placebo comparator.
  Arms: Thunderbeat™
Device: Standard of care scissors, ligatures, clips, and sutures
  Arms: Control Group

SUMMARY:
The Whipple procedure is the standard method for therapy for cancerous tumors, inflammation, and stenosis (narrowing) near the head of the pancreas. This is a prospective study to assess whether or not use of the Thunderbeat™ device may decrease blood loss and postoperative morbidity (the presence of illness or disease). The findings will then be compared to patients whose Whipple procedure will be performed using conventional dissection and hemostasis techniques.

DETAILED DESCRIPTION:
As the pancreas is fed by many vessels, it is necessary to use lots of ligatures, clips and sutures for hemostasis after dissection. This dissection technique is very time consuming and requires numerous changes of instruments. The devices the investigators currently have available for use in the operating suite are EnSeal and LigaSure. A new type of surgical scissors that delivers ultrasonically generated frictional heat energy and electrically generated bipolar energy simultaneously, known as the Thunderbeat™ (Olympus, Japan), is now an available alternative for dissection and hemostasis.

Thunderbeat™ was provided FDA clearance in March 2012 for use in open, laparoscopic, and endoscopic surgery, or in any procedure in which cutting, vessel ligation (sealing and cutting), coagulation, grasping and dissection is performed.

The Thunderbeat™ device provides the first integration of both bipolar and ultrasonic energies delivered simultaneously from a single multi-functional instrument. This integration provides the surgeon the ability to rapidly cut tissue with ultrasonic energy and to create reliable vessel seals with bipolar energy without having to change devices. The current is provided by a special generator and contains a very high capacity with a low voltage. The body's proteins, such as collagen and elastin, are converted so a permanently sealed zone results. As the tissue between the branches is sealed, lateral thermic tissue damages can be limited to a minimum. Several authors have described a tendency of reduced intraoperative blood loss with bipolar energy devices. Other trials show reduced operating time when a bipolar device is utilized in several surgical procedures, such as thyroid, hepatic, urologic, hemorrhoidectomy and gynecology surgery.

Correct dissection in the operating field is very important to avert secondary bleeding or other complications, which might cause re-operation or elevate the patients' morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo an elective open or laparoscopic Whipple procedure
* At least 22 years of age.
* Karnofsky performance status greater than or equal to 80%.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Surgeon's opinion at the time of dissection that the subject's well being (e.g. bleeding or other independent acute health problems) would be compromised.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hawkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 01/01/2015 and closed to participant enrollment on 08/09/2017.
Pre-assignment Details: There were 44 enrolled to the study. 12 were enrolled but were not randomized to an arm and did not start the study due to reasons such as ineligibility, physician discretion, and because the Thunderbeat was not in the operating room.
Groups:
- Thunderbeat™: * In the Thunderbeat™ group, dissection and hemostasis of vessels will be performed using the Thunderbeat™ device (Olympus, Japan).
  * Thunderbeat uses ultrasonic and high frequency bipolar energy simultaneously to seal and cut tissue compared to placebo comparator.
Period: Overall Study
Arm/Group | Control Group | Thunderbeat™
Started | 13 | 19
Completed | 13 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Thunderbeat™ | Total
Number analyzed (Participants) | 13 | 19 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.9) | 64.8 (11.3) | 64.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 18 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 19 | 32
Received Neoadjuvant Therapy [Count of Participants; unit: Participants] | 3 | 5 | 8
Body Mass Index (BMI) > 30 kg/m^2 [Count of Participants; unit: Participants] | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Operative Blood Loss
Description: * The measurement of estimated blood loss (EBL) will come from the intraoperative anesthesia notes where (EBL) is recorded during each surgical procedure
  * The estimate of operative blood loss is measured by volume in the suction canisters and pads and is historically documented by the operative nursing staff during the operation.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
mL | 263.5 (190.0) | 480.2 (300.5)
Statistical Analysis 1: Comparison: Control Group vs Thunderbeat™; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Post-op Morbidity
Description: -This is a prospective study to evaluate post-operative morbidity following use of the ThunderbeatTM device during the Whipple procedure. This will be compared to patients whose Whipple procedure will be performed using conventional dissection and hemostasis techniques.
Time Frame: Up to 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
Participants | 7 | 8
Statistical Analysis 1: Comparison: Control Group vs Thunderbeat™; Test type: Superiority; p = 0.513, Chi-squared

3. Secondary Outcome: Operative Time
Description: -Operation time measured from the beginning of the surgical procedure (incision of the skin) to the end of the surgical procedure (closure of the skin).
Time Frame: Day of surgery
Measure: Median (Full Range); unit: minutes
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
minutes | 220 [143 to 296] | 270 [183 to 491]

4. Secondary Outcome: Cost Using Thunderbeat Device
Description: -Calculated by the indirect and direct costs during the hospital stay and the costs accumulated 90 days postoperatively
Time Frame: Up to 90 days postoperatively
Population: The data for this outcome measure was not collected.
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Anesthesia Time
Description: -Anesthesia time measured from the initiation of anesthesia induction to the time of extubation
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
minutes | 282.7 (50.8) | 357.3 (89.2)
Statistical Analysis 1: Comparison: Control Group vs Thunderbeat™; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants Who Experienced Perioperative Complications
Description: -Complications experienced during surgery will be reviewed including:
  * Iatrogenic injury
  * need for conversion from laparoscopic approach to open procedure
  * need for the use of other hemostatic devices or therapies
  * intraoperative requirement of blood product transfusion
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
Participants | 0 | 3
Statistical Analysis 1: Comparison: Control Group vs Thunderbeat™; Test type: Superiority; p = 0.132, Chi-squared

7. Secondary Outcome: Number of Participants Who Experienced Postoperative Complications
Description: -Complications experienced after surgery will be reviewed including:
  * secondary bleeding/hematoma
  * wound infection
  * gastroparesis
  * postoperative pancreatic fistula
  * intraabdominal abscess
  * anastomotic leakage
  * re-intervention (operational)
  * postop requirement for blood product transfusion
  * hospital mortality
Time Frame: Up to 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Thunderbeat™
Number analyzed (Participants) | 13 | 19
Participants
  Readmission | 2 | 3
  Mortality | 0 | 0
  Bleeding/hematoma | 0 | 0
  Wound infection | 0 | 1
  Gastroparesis | 2 | 3
  Pancreatic fistula | 0 | 1
  Intraabdominal abscess | 0 | 1
  Anastomotic leakage | 0 | 1
  Blood product transfusion (anemia) | 1 | 0
Statistical Analysis 1: Comparison: Control Group vs Thunderbeat™; Statistical analysis #1 is for readmission; Test type: Superiority; p = 0.975, Chi-squared
Statistical Analysis 2: Comparison: Control Group vs Thunderbeat™; Statistical analysis #2 is for wound infection; Test type: Superiority; p = 0.401, Chi-squared
Statistical Analysis 3: Comparison: Control Group vs Thunderbeat™; Statistical analysis #3 is for gastroparesis; Test type: Superiority; p = 0.975, Chi-squared
Statistical Analysis 4: Comparison: Control Group vs Thunderbeat™; Statistical analysis #4 is for pancreatic fistula; Test type: Superiority; p = 0.401, Chi-squared
Statistical Analysis 5: Comparison: Control Group vs Thunderbeat™; Statistical analysis #5 is for intraabdominal abscess; Test type: Superiority; p = 0.219, Chi-squared
Statistical Analysis 6: Comparison: Control Group vs Thunderbeat™; Statistical analysis #6 is for anastomotic leakage; Test type: Superiority; p = 0.401, Chi-squared
Statistical Analysis 7: Comparison: Control Group vs Thunderbeat™; Statistical analysis #7 is for blood product transfusion (anemia); Test type: Superiority; p = 0.219, Chi-squared

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from the time of surgery through 90 days following completion of surgery.
Description: -Surgical complications will not be considered adverse events associated with the study, unless unanticipated and possibly related to the use of the Thunderbeat device.
Arm/Group | Control Group | Thunderbeat™
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/19
Other Adverse Events (participants affected / at risk) | 0/13 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT02204124/Prot_SAP_000.pdf